CLINICAL TRIAL: NCT05851846
Title: Amygdala Insula Retraining in the Management of Long COVID Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leonardo Tamariz, Staff physician, Miami VA Healthcare System
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1677529-1
Record Dates: First submitted 2023-05-08; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: What list of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mind body intervention + Usual care: The intervention will be delivered virtually
  Interventions: Behavioral: Amygdala insula retraining
- Control arm (No Intervention): The participants in the comparator group will be wait listed for the intervention

INTERVENTIONS:
Behavioral: Amygdala insula retraining — Mind body intrevention
  Arms: Intervention

SUMMARY:
The goal of the study is to compare a mind body intervention against usual care in patients with fatigue with long COVID.

Our research questions include

1. Is the mind body intervention additive to usual care in long COVID
2. Can the mind body intervention change laboratory markers, heart rate variability and dysautonomia.

DETAILED DESCRIPTION:
More than 30 percent of the over 70 million individuals in the United States who experienced an acute COVID-19 infection as a result of severe acute respiratory coronavirus-2 (SARS-CoV2), have variety of lingering and disabling symptoms that last beyond the acute phase of the illness. [1]This condition is referred to as Post-Acute Sequalae SARS-CoV-2 infection (PASC). Symptoms (including fatigue, post-exertional malaise (PEM), cardiovascular dysfunction, respiratory distress, gastrointestinal disturbances, and dermatologic issues) associated with PASC vary and can affect multiple organ systems. These symptoms are similar to, in extent and degree, to other neuro-immune conditions such as Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). PASC, as with ME/CFS, is likely to pose a significant impact on the healthcare system and patient's quality of life. An unmet need exists as the susceptibility and pathogenesis of PASC remains yet to be fully elucidated. Emerging evidence suggests that existing interventions widely used for other neuro-immune conditions may prove equally effective in the treatment of PASC. Repurposing of drugs or identification of new drugs will take time. Still, there is growing evidence of the mind-body connection in modulating the autonomic, central and peripheral nervous systems as well as the immune system and the gastrointestinal tract. Recent studies have documented that holistic strategies such as mindfulness, meditation, and amygdala and insula retraining (AIR) have an objective measurable effect on heart rate variability, fatigue, pain, quality of life, depression, anxiety, and gastrointestinal symptoms. The mechanisms proposed include activation of vagus nerve, balancing the autonomic nervous system, reducing stress, and improving immune function. AIR is based on the principle that viral, bacterial, or environmental insults can sensitize the amygdala, which becomes hypervigilant and unleashes a cascade of hormonal responses that perpetuate a state of neuroinflammation and dysautonomia. AIR de-sensitizes the amygdala, breaking vicious cycles and reducing the maladaptive release of hormones and cytokines. Our clinical group has already recommended the use of AIR with great anecdotical response in clinical practice. This strategy is readily available and has no contraindications or risks. We aim to conduct a pilot study of AIR to generate preliminary data for a larger, federally funded trial. Our specific aims are:

1. Identify 130 subjects within the Miami Veteran's Administration (VA) Medical Center who experienced an acute COVID-19 infection and continue to experience persistent moderate fatigue (using standard questionnaires). Subjects will be randomized to either 1. AIR + standard of care or 2. Standard of care/wait list. Individuals in this latter arm will be waitlisted to receive the AIR intervention after they complete the study.
2. Collect standard questionnaires recommended by the Veterans Affairs Healthcare System at baseline, three, and six months to capture levels of fatigue (primary outcome), post exertional malaise (PEM), brain fog, pain, and other symptoms and compare changes over time across the two study arms.
3. Collect objective biometric data in a sample of patients at baseline and at three and six months to explore potential mediating mechanisms: heart rate variability, heart rate and blood pressure sitting and standing, inflammatory markers (c-reactive protein, cortisol, and Epstein Barr viral reactivation. The laboratory tests will not be collected for research purposes as they are collected for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be:

  1. Fulfill the definition of PASC
  2. Be a patient in the Miami VA post COVID clinic
  3. Have access to a computer or phone
  4. Report moderate fatigue as defined by the clinically obtained surveys in the post COVID clinic. The rationale for this inclusion criteria is that 85% of our post COVID patient report fatigue and fatigue is a target outcome can be followed.
  5. A probable or confirmed diagnosis of acute COVID-19 infection as per WHO guidelines.
  6. Have no evidence of cardiac or pulmonary end organ damage, as per WHO definition. We will define not having end organ damage as a normal ejection fraction on echocardiogram and no pulmonary infiltrates on a non-contrast computed tomography (CT) of the chest during the work-up of the long COVID clinic.

Exclusion Criteria:

* There will be no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Modified Yorkshire COVID-19 scale | 3 months
  Long COVID symptom scale

SECONDARY OUTCOMES:
Heart rate variability | 3 months
  SSDN
COMPASS-31 | 3 months
  Dysautonomia scale

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Institute for Neuroimmune Medcince, Fort Lauderdale, Florida
  - Miami VAHS, Miami, Florida
  - Institute for Neuroinmune medicine, Miami, Florida